CLINICAL TRIAL: NCT05979558
Title: Study of Caudal Ropivacaine With or Without Dexmedetomidine for Postoperative Analgesia in Pediatric Infra-umbilical Surgery: A Double-blinded Randomized Control Trial
Brief Title: Caudal Ropivacaine With or Without Dexmedetomidine for Post Operative Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Academy of Medical Sciences, Nepal (Other Government)
Responsible Party: Principal Investigator, Kaushal Tamang, Principal Investigator, National Academy of Medical Sciences, Nepal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NamsNepal
Record Dates: First submitted 2023-07-21; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Ropivacaine; Infraumbilical Surgery; Dexmedetomidine; Analgesia
Keywords: ropivacaine; caudal ropivacaine; dexmedetomidine; placebo; analgesia; infraumbilical surgery
MeSH Terms: conditions — Agnosia | interventions — Ropivacaine; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Children were randomly assigned to two groups having 31 children in each, by using a computer-generated table of random numbers which was enclosed in a sealed envelope and was opened by an anesthesiologist who were not involved in the study.
Who Masked: Participant, Care Provider
Masking Description: Children were randomly assigned to two groups having 31 children in each, by using a computer-generated table of random numbers which was enclosed in a sealed envelope and was opened by an anesthesiologist who were not involved in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ropivacaine with dexmedetomidine (Experimental)
  Interventions: Drug: ropivacaine with dexmedetomidine
- Ropivacaine with Normal Saline (Placebo Comparator)
  Interventions: Drug: Ropivacaine with placebo

INTERVENTIONS:
Drug: ropivacaine with dexmedetomidine — this group received with ropivacaine with dexmedetomidine
  Arms: Ropivacaine with dexmedetomidine
Drug: Ropivacaine with placebo — this group received with ropivacaine with normal saline
  Arms: Ropivacaine with Normal Saline

SUMMARY:
The goal of this clinical trial is to evaluate the postoperative analgesic effects of caudal Ropivacaine with or without Dexmedetomidine in pediatric infraumbilical surgery. The main question[s] it aims to answer are:

• if Caudal Dexmedetomidine with Ropivacaine would prolong the duration of analgesia in children undergoing infraumbilical surgery.

Participants will receive ropivacaine with dexmedetomidine in infraumbilical surgery.

If there is a comparison group: Investigators will compare this with ropivacaine with a placebo to see if the duration of analgesia differs.

DETAILED DESCRIPTION:
Children have significant pain following surgery. It has been under-managed most of the time. Poorly controlled post-operative pain increases the morbidity. It leads to post-operative agitation, urinary retention, nausea and vomiting, hypoxia, pulmonary edema, cardiovascular and temperature instability. So, postoperative pain management is an essential and important component of pediatric postoperative care. Adequate pain control after surgery permits early mobilization, reduces postoperative complication, prevents development of fear and anxiety and allows early hospital discharge.

Caudal block is one of the modality of multimodal analgesia. It is a well-established, effective and relatively safe technique used for intra and post-operative analgesia in children undergoing abdominal and lower limb surgery. It provides excellent analgesia, reduces intra-operative anesthetics drug requirements, ensures pain free recovery from anesthesia, decreases stress response and avoids deleterious adverse effects of narcotic drugs.

However, the main disadvantage of caudal block is being its short duration of action with sole local anesthetics. Even long-acting local anesthetic drugs such as bupivacaine provides only 4-8 hours of analgesia. The insertion of catheter in caudal space to administer repeated doses or continuous infusions of local anesthetic drug is not popular because of concerns of infection. So, various adjuvants like Fentanyl, Morphine, Ketamine, clonidine, Dexmeditomidine etc. have been used to prolong the duration of analgesia.

Morphine and Fentanyl are opioids that have been used traditionally in combination with a local anesthetic to achieve prolonged anesthetic effect. The addition of opioid does provide better analgesia but there is a possibility of an increased incidence of pruritus, urinary retention, nausea, vomiting and respiratory depression. Similarly, Ketamine and Clonidine are the widely preferred adjuvant to caudal block but have their own number of unpleasant adverse effects8.

Hence, there is still ongoing investigations to find for an adjuvant that can safely prolong caudal analgesia. Recently, Dexmedetomidine has been used for this purpose. Various studies have described the use of Dexmedetomidine with local anesthetic drugs in caudal block for the management of postoperative pain in children. Saadawy et al. found that 1μg/kg caudal dexmedetomidine with bupivacaine was associated with an extended duration of postoperative analgesia while in other studies 2μg/kg Dexmedetomidine was used with caudal Bupivacaine or Ropivacaine for providing postoperative analgesia in children undergoing lower abdominal and perineal surgeries.

Dexmedetomidine is a highly specific and selective α2-adrenoceptor agonist that has been described as a safe and effective additive in many anesthetic procedures. In contrast to other agents, it has a sympatholytic, analgesic and sedative effects. It is remarkably free from side effects except for hypotension and bradycardia. But studies investigating its analgesic property in our population are limited.

Ropivacaine is a long-acting amino amide local anesthetic drug and was the first to be formulated as a pure S-enantiomer. It is reported to have a better safety profile than Bupivacaine with less risk for central nervous system and cardiac toxicity 10. It also decreases unwanted motor block than Bupivacaine, which makes it a more suitable agent for caudal epidural analgesia6.

Dexmedetomidine with Ropivacaine is commonly used to prolong the caudal analgesia in western population but have not been well studied in our pediatric population. So investigators designed this study to determine analgesic effect of caudal Dexmedetomidine with Ropivacaine in pediatric infraumbilical surgeries.

HYPOTHESIS Caudal Dexmedetomidine with Ropivacaine would not prolong the duration of analgesia in children undergoing infraumbilical surgery.

GENERAL OBJECTIVES To evaluate the postoperative analgesic effects of caudal Ropivacaine with or without Dexmedetomidine in pediatric infraumbilical surgery SPECIFIC OBJECTIVES

1. To compare rFLACC score (revised Face, Legs, Activity, Cry, and Consolability)in 24 hours of postoperative period.
2. To compare the time for first rescue analgesia.
3. To evaluate the total analgesics consumption in 24 hours of postoperative period.
4. To observe the side effects of study drugs (vomiting and bradycardia).

ELIGIBILITY:
Inclusion Criteria:

* Children of either sex aged 2-7 years
* ASA (American Society of Anesthesiologist) physical status I or II
* Patients undergoing elective infraumbilical surgeries

Exclusion Criteria:

* History of neuromuscular or psychiatric disease
* Coagulation disorders
* Skin lesion at the site of injection
* Spine deformity
* History of developmental delay
* Allergy to study drugs

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Duration of analgesia: | upto first 24 hour after intervention
  The primary outcome will be the duration of analgesia defined as the time period between administration of study drugs to first need of rescue analgesia when until the time of rFLACC score (revised Face, Legs, Activity, Cry, and Consolability) reached ≥4.
Post-operative pain Assessment (rFLACC score) rFLACC score (revised Face, Legs, Activity, Cry, and Consolability) | first 24 hour after intervention
  Each of the five categories F (face), L (legs), A (Activity), C (Cry), C (Consolability) will be scored from 0 to 2 which results total score in between zero and ten.
Total analgesics consumption in first 24 hours postoperative period | first 24 hours after intervention
  If r-FLACC pain score ≥4 at any time, an injection Paracetamol 15mg/kg will be given. If the r-FLACC pain score still ≥4 after 30 minutes of injection Paracetamol, then the child will treated with an injection Pethidine 0.5mg/kg. After that, an injection Paracetamol at 15mg/kg will be given 6 hourly. Total analgesic consumption in the first 24 hours will be calculated by adding the total analgesic consumed in 24 hours after the intervention.

SECONDARY OUTCOMES:
Side effects of study drugs | monitored for 24 hours and treated accordingly
  Adverse events such as nausea, vomiting, bradycardia, respiratory depression and urinary retention will be monitored for 24 hours and treated accordingly

CONTACTS AND LOCATIONS:
Overall Officials: Kaushal Tamang, MBBS,MD, Principal Investigator — NAMS; Bidur K Baral, MBBS,MD, Study Chair — NAMS; Sadichhya S Malla, MBBS,MD, Study Chair — Kanti Hospital
Locations (1):
- National Academy of Medical Sciences (NAMS), Kathmandu, Bagmati, Nepal